CLINICAL TRIAL: NCT06848179
Title: Smartphone-Based Use of Phonocardiography Technique for Estimating Heart Rate and Heart Rate Variability: Performance Study
Status: Not yet recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Laboratory of Data Discovery for Health (Unknown)
Responsible Party: Principal Investigator, Dr. Joshua Wing-Kei Ho, Associate Professor, The University of Hong Kong
Other Study IDs: AUSC-HR
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Exercise
Keywords: Auscultation; Smartphone; Heart Sounds; Heart Auscultation; Phonocariodgraphy
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy Participants: Participants deemed ready for physical activity by the Physical Activity Readiness Questionnaire (PAR-Q)
  Interventions: Diagnostic Test: Computer algorithms; Behavioral: Exercise

INTERVENTIONS:
Diagnostic Test: Computer algorithms — Collection of computer algorithms called ausculto® that is designed to perform heart sound analysis to estimate heart rate and heart rate variability
  Other Names: ausculto®; Vitogram®
Behavioral: Exercise — Participants will be requested to exercise to raise their HR over the resting range while heart-related physiological signals are collected.

SUMMARY:
This study aims to investigate the use of heart sound recordings, or phonocardiograms, recorded with smartphones' built-in microphones and accessory microphones to estimate heart rate (HR) and heart rate variability (HRV). HR refers to the number of heart beats per minute, while HRV refers to the variation in the intervals between heart beats.

Participants will have their heart sounds (phonocardiograms) recorded before and after exercise, and electrocardiogram (ECG) and photoplethysmogram (PPG) data recorded before, during, and after exercise to induce a wide range of HR.

Researchers will match the phonocardiograms, ECG, and PPG data to create a database for use in future training and testing of algorithms (including artificial intelligence (AI)).

ELIGIBILITY:
Inclusion Criteria:

* With no tattoos on their body where a smartwatch will be placed

Exclusion Criteria:

* Not ready to undertake physical activity as assessed by the Physical Activity Readiness Questionnaire (PAR-Q) derived from the Canadian Society for Exercise Physiology
* Implanted active medical devices in the torso, such as pacemakers and defibrillators
* Failure to collect baseline heart sound time series from ECG or both smartphone and auscultation pin before exercise

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Apparently healthy volunteers aged 18-69 recruited from the general public
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
HR estimation | Day 0
  The algorithm will estimate participants' HR from phonocardiograms at multiple timepoints. The concordance correlation coefficient, mean bias, and limits of agreement will be calculated for HR with ECG-derived HR as the gold standard.
HRV estimation | Day 0
  The algorithm will estimate participants' HRV from phonocardiograms at multiple timepoints. The absolute difference (error) in HRV estimation will be calculated with ECG-derived HRV as the gold standard.

SECONDARY OUTCOMES:
Participants' comfort level for devices used in this study | Day 0
  A survey will be given to participants after heart data collection to evaluate their preferences and comfort level when using the different devices to measure HR and HRV.

IPD SHARING:
Plan to Share IPD: No